CLINICAL TRIAL: NCT00477971
Title: Phase III Trial of Stem Cell Transplantation Compared to Parenteral Melphalan and Oral Dexamethasone in the Treatment of Primary Systemic Amyloidosis (AL)
Brief Title: Low-Dose Melphalan and Dexamethasone Compared With High-Dose Melphalan Followed By Autologous Stem Cell Transplant in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546745; P30CA015083 (NIH); MC0482 (Other: Mayo Clinic Cancer Center); 1691-05 (Other: Mayo Clinic IRB); NCI-2009-01329 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Dexamethasone; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Patients receive low-dose melphalan IV over 15-30 minutes on day
  1 or orally once daily on days 1-7 and oral dexamethasone on days 1-4 and 22-25. Treatment repeats every 6 weeks for 10 courses.
  Study treatment beyond one year is not allowed.
  Interventions: Drug: dexamethasone; Drug: melphalan
- Arm B (Experimental): Patients receive filgrastim (G-CSF) on days -7 to -3 and undergo autologous hematopoietic stem cell (HSC) collection. Patients receive high-dose melphalan IV over 1 hour on days -2 and -1 and undergo autologous HSC transplantation on day 0.
  Interventions: Biological: filgrastim; Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — No administration information given
  Arms: Arm B
Drug: dexamethasone — Given orally
  Arms: Arm A
Drug: melphalan — Given IV or orally
Procedure: autologous hematopoietic stem cell transplantation — Given on day 0
  Arms: Arm B

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan and dexamethasone, work in different ways to stop the growth of plasma cells, either by killing the cells or by stopping them from dividing. Having an autologous stem cell transplant to replace the blood-forming cells destroyed by chemotherapy, allows higher doses of chemotherapy to be given so that more plasma cells are killed. By reducing the number of plasma cells, the disease may progress more slowly. It is not yet known whether combination chemotherapy is more effective than chemotherapy followed by an autologous stem cell transplant in treating primary systemic amyloidosis.

PURPOSE: This randomized phase III trial is studying the side effects and how well giving low-dose melphalan together with dexamethasone works compared with high-dose melphalan followed by an autologous stem cell transplant in treating patients with primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare hematologic response rate in patients with primary systemic amyloidosis treated with conventional chemotherapy comprising low-dose melphalan and dexamethasone vs high-dose melphalan followed by autologous stem cell transplantation.
* Compare the toxicity of these regimens in these patients.

Secondary

* Compare the overall and progression-free survival of patients treated with these regimens.
* Compare the regression of organ involvement in patients treated with these regimens.
* Compare the duration of response in patients treated with these regimens.
* Correlate clonal burden and time to in vitro amyloid formation with clinical outcomes in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Compare the information-seeking behavior in patients treated with these regimens.

OUTLINE: This is a comprehensive cohort study comprising a randomized option and a nonrandomized option. Patients consenting to randomization are stratified by risk group (high vs low) and ECOG performance status (0-1 vs 2). They are then randomized to 1 of 2 treatment arms. Patients not consenting to randomization choose their treatment arm.

* Arm I: Patients receive low-dose melphalan IV over 15-30 minutes on day 1 or orally once daily on days 1-7 and oral dexamethasone on days 1-4 and 22-25. Treatment repeats every 6 weeks for 10 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive filgrastim (G-CSF) on days -7 to -3 and undergo autologous hematopoietic stem cell (HSC) collection. Patients receive high-dose melphalan IV over 1 hour on days -2 and -1 and undergo autologous HSC transplantation on day 0.

Blood and bone marrow samples are collected at baseline. Samples are examined by PCR, cDNA, and nucleotide sequence analysis to determine VH and VL gene families and carrier status. Urine is collected at baseline and analyzed for light-chain protein levels by exclusion chromatography.

Quality of life is assessed at baseline, at months 3, 9, and 12, at completion of study treatment, and then every 6 months for up to 5 years.

After completion of study treatment, patients are followed every 6 months for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary systemic amyloidosis

  * Amyloid light-chain (AL) disease
* Monoclonal protein by immunoelectrophoresis or immunofixation of the serum or urine OR abnormal free light-chain ratio
* The following amyloid syndromes* are allowed:

  * Amyloid hepatomegaly
  * Cardiomyopathy
  * Proteinuria
  * Peripheral or autonomic neuropathy
  * Soft tissue involvement including the tongue, submandibular tissues, and vascular claudication
  * Diffuse interstitial pulmonary AL disease allowed if pulmonary function is adequate to allow safe transplantation NOTE: *Presence of amyloid deposits in a plasmacytoma or in bone marrow vessels in an asymptomatic patient does not constitute an amyloid syndrome
* No secondary or familial amyloidosis
* No multiple myeloma with lytic or destructive bone lesions or myeloma cast nephropathy
* No multiple myeloma with > 30% plasma cells in the bone marrow
* No amyloidosis manifested only by carpal tunnel syndrome or purpura

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 6 times ULN
* Creatinine ≤ 3.0 mg/dL
* No NYHA class IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* Prior alkylating agents, immunosuppressive drugs, or steroids allowed provided they were given for < 1 month

  * Therapeutic steroid doses of ≤ 15 mg per day (or equivalent) allowed at discretion of physician
* No concurrent participation in another clinical trial involving a pharmacologic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-10; Primary Completion 2012-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morie A. Gertz, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2005 to August 2012, 89 participants were recruited.
Pre-assignment Details: This study was originally designed as a randomized Phase III clinical trial; however the unwillingness of participants to be randomized to treatment led to changes. The protocol was amended to allow participants to choose between the two regimens.
Groups:
- Low-Dose Melphalan: Patients receive low-dose melphalan 20 mg/m^2 IV over 15-30 minutes on day 1 or 0.12 mg/kg tablet orally once daily on days 1-7 and dexamethasone 40 mg orally on days 1-4 and 22-25. Treatment repeats every 6 weeks for 10 courses. (Study treatment beyond one year is not allowed.)
- High-Dose Melphalan + Autologous HSC: Patients receive filgrastim (G-CSF) 10 mg/kg/day on days -7 to -3 and undergo autologous hematopoietic stem cell (HSC) collection. Patients receive high-dose melphalan 140 mg/m^2 IV for low risk or 200 mg/m^2 IV for high risk patients over 1 hour on days -2 and -1 and undergo autologous HSC transplantation on day 0.
Period: Overall Study
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC
Started | 34 | 55
Completed | 17 | 49
Not Completed | 17 | 6
Not completed — Disease progression | 6 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Death | 2 | 4
Not completed — Alternative treatment | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC | Total
Number analyzed (Participants) | 34 | 55 | 89
Age, Continuous [Median (Full Range); unit: years] | 62 [48 to 74] | 57 [44 to 73] | 59 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 17 | 39 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 32 | 51 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 34 | 55 | 89
ECOG Performance Score [Number; unit: participants] — Classifies patients according to their functional impairment. 0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  participants
    0-1 | 25 | 50 | 75
    2 | 9 | 5 | 14
Risk Group [Number; unit: participants] — Low Risk (requires all of the following): 1 or 2 organs involved, Cardiac EF >= 50%, Age <= 65 years, NYHA class 1 or 2, Alkaline phosphatase <= 4 x institutional ULN, cardiac involvement fully compensated or asymptomatic, serum creatinine <= 2.0 mg/dL
  High Risk (any one of the following): >2 organs involved, Cardiac EF <50%, Age > 65 years, NYHA class 3, Alkaline phosphatase 4-6 x institutional ULN, symptomatic cardiac involvement, serum creatinine 2.1-3.0 mg/dL
  participants
    Low | 20 | 38 | 58
    High | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate
Description: Response that was confirmed on 2 consecutive evaluations during treatment. A hematologic response consisted of a Complete response, Very Good Partial Response or Partial Response.
  * Complete Response (CR): Complete disappearance of M-protein from serum and urine on immunofixation, normalization of Free Light Chain (FLC) ratio and <5% plasma cells in bone marrow.
  * Very Good Partial Response (VGPR): >=90% reduction in serum M-component; Urine M-Component <=100 mg per 24 hours.
  * Partial Response (PR): >=50% reduction in serum M-component and/or Urine M-Component >=90% reduction or <200 mg per 24 hours; or >=50% decrease in difference between involved and uninvolved FLC levels.
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC
Number analyzed (Participants) | 34 | 55
percentage of participants | 55.9 [37.9 to 72.8] | 69.1 [55.2 to 80.9]

2. Secondary Outcome: 3 Year Overall Survival
Description: Percentage of patients who were alive at 3 years. The 3-year survival rate was estimated using the Kaplan Meier method.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC
Number analyzed (Participants) | 34 | 55
percentage of participants | 58.8 [44.4 to 77.9] | 83.6 [74.7 to 94]

3. Secondary Outcome: Organ Response to Treatment
Description: Organ response was evaluated on the basis of improvement of one or more affected organ; only one parameter was required to satisfy the criteria. Response needed to be maintained for a minimum of 3 months to be considered valid.
  Renal response required a 50% reduction in 24-hour urine protein excretion (at least 0.5 g/d) with stable creatinine. Cardiac response required one of >= 2-mm reduction in the interventricular septal (IVS) thickness by echocardiogram, or improvement of ejection fraction by >= 20%, or improvement by 2 NYHA classes without an increase in diuretic use. Hepatic response required either >= 50% decrease in (or normalization of) an initially elevated alkaline phosphatase level or reduction in the size of the liver by at least 2 cm by radiographic determination. Gastrointestinal tract improvement was defined as normalization of a low serum carotene level, or reduction of diarrhea to < 50% of previous movements/day, or decrease in fecal fat excretion by 50%.
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC
Number analyzed (Participants) | 34 | 55
percentage of participants | 26.5 [12.8 to 44.4] | 29.1 [17.6 to 42.9]

4. Post Hoc Outcome: 3-Year Progression Free Survival
Description: Percentage of patients who were progression free at 3 years. The 3-year progression free rate was estimated using the Kaplan Meier method.
  Progression is assessed when one of the following occur:
  * reappearance of monoclonal protein by immunofixation,
  * Increase in serum monoclonal paraprotein to >25% above the lowest response level,
  * Increase in urine M-protein to > 25% above the lowest remission value for 24-hour excretion.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC
Number analyzed (Participants) | 34 | 55
percentage of participants | 29.1 [17.2 to 49.4] | 51.7 [39.8 to 67]

ADVERSE EVENTS:
Arm/Group | Low-Dose Melphalan | High-Dose Melphalan + Autologous HSC
Serious Adverse Events (participants affected / at risk) | 6/34 | 3/55
Other Adverse Events (participants affected / at risk) | 34/34 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Melphalan (N=34) | High-Dose Melphalan + Autologous HSC (N=55)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Melphalan (N=34) | High-Dose Melphalan + Autologous HSC (N=55)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 32 (33)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (41) | 49 (63)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 5 (7)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 25 (27)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 12 (12)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 32 (35)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 17 (19)
Chest pain (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 32 (140) | 48 (140)
Fatigue (General disorders) | 33 (178) | 55 (197)
Fever (General disorders) | 1 (1) | 8 (8)
General symptom (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (4) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 3 (5) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious meningitis (Infections and infestations) | 0 (0) | 1 (1)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (7) | 4 (5)
Sepsis (Infections and infestations) | 2 (2) | 10 (12)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 4 (4) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative gastrointestinal injury - Appendix (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative hepatobiliary injury - Gallbladder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (5)
Alkaline phosphatase increased (Investigations) | 2 (2) | 10 (11)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 9 (10)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 6 (15) | 21 (33)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 9 (20) | 51 (56)
Lymphocyte count decreased (Investigations) | 2 (4) | 3 (5)
Neutrophil count decreased (Investigations) | 8 (18) | 52 (60)
Platelet count decreased (Investigations) | 10 (27) | 52 (65)
Weight loss (Investigations) | 13 (24) | 21 (26)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 31 (34)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 9 (12)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 11 (11)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 19 (72) | 21 (60)
Syncope (Nervous system disorders) | 3 (6) | 4 (6)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 4 (4)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal failure (Renal and urinary disorders) | 4 (5) | 4 (5)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 11 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 33 (34)
Thrombosis (Vascular disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes